CLINICAL TRIAL: NCT01443273
Title: Thrombophilic Risk Factors in Preterm and Infants Treated at Ha'Emek Medical Center Between the Years 1990 to 2010
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit and, HaEmek Medical Center, Israel
Other Study IDs: 0041-11-EMC
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Premature; Thrombosis
Keywords: Newborns
MeSH Terms: conditions — Premature Birth; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with thrombotic events: All infants (premature and term) diagnosed at the Neonatal Intensive Care Unit with thrombotic events
  Interventions: Other: Medical Records study

INTERVENTIONS:
Other: Medical Records study — No interventions will be done related to the study besides summary of the Medical Files.

SUMMARY:
There are several factor that can be related to Neonatal Thrombotic events. Among them hypercoagulability can be the cause of those events. Factor V Leiden (FVL) and Prothrombin mutation are the most common causes of hereditary thrombophilia. The incidence of in the arab population is known to be higher than the incidence in another western populations. The purpose of this study is to review retrospectively the thrombophilic risk factors that were found in a cohort of premature babies and term newborns treated and investigated at the Neonatal Intensive Care Unit and at the Pediatric Hematology Unit.

DETAILED DESCRIPTION:
All the demographic and clinical data will be summarized. Factors non related to the coagulation system like catheters, severe infections or congenital heart defects will be recorded. Also a full workup of prothrombotic risk factors are routinely performed in those infants. The study included basic coagulation analysis, Protein C, S and Antithrombin III activity, Activated Protein C Resistance, serum homocystein, lipoprotein (a) and Lupus Anticoagulant.

Also the three common genetic factors are analysed including Factor F Leiden (G1691A), Prothrombin Mutation (G20210A) and MTHFR polymorphism (C677T).

ELIGIBILITY:
Inclusion Criteria:

-All newborns (Term and Premature) diagnosed with Neonatal Thrombotic events between year 1990 to 2010.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns (Term and Premature) diagnosed with Neonatal Thrombotic events between year 1990 to 2010.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The frequency of thrombophilic risk factors in preterms and infants | One year
  Recruitment of all premature and term infants born at Emek Medical Center and suffer from thrombotic events.

CONTACTS AND LOCATIONS:
Overall Officials: Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel